CLINICAL TRIAL: NCT06834815
Title: Effect of Probiotics on Chromogenic Bacteria and Extrinsic Stains in Children
Brief Title: Investigating the Bactericidal Effect of Probiotics on Chromogenic Bacteria in Children An In Vivo and In Vitro Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-Rec IR102420
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-11

CONDITIONS: Black Stains
Keywords: probiotics; chromogenic bacteria; black stains
MeSH Terms: interventions — Probiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: probiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- before and after probiotic administration (Experimental): all patients will submit an unstimulated salivary sample of 1ml will in sealed test tube
  * then the patients will receive probiotics for 14 days .
  * after 14 days and another salivary sample will be collected
  Interventions: Drug: Probiotic with Prebiotic

INTERVENTIONS:
Drug: Probiotic with Prebiotic — After assigning the patients , all patients will submit an unstimulated salivary sample of 1ml will in sealed test tubes then stored in a deep freezer until microbiological evaluation, then they'll receive an oral prophylaxis session.
  * The patients will receive probiotics for 14 days given to them in a sealed box.
  * All patients will be followed up after 14 days and another salivary sample will be collected and sent for microbiological assessment.

SUMMARY:
To investigate the bactericidal effect of probiotics (Streptococcus salivarius M18 and Lactobacillus reuteri) on two types of bacteria (Aggregatibacter actinomycetemcomitans and Actinomyces naeslundii) causing black stains of teeth in vitro.

DETAILED DESCRIPTION:
In vitro:

An unstimulated salivary sample will be taken from patients having black stains. The two types of bacteria of each condition will be cultured, amplified, and measured in the laboratory from the saliva of these patients. After that, one type of probiotics will be applied to these bacteria separately and the same bacterial measurement will be done to evaluate the bactericidal effect of the probiotics on these bacteria, aiming to find the minimal inhibitory concentration of the probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with black stains on teeth scored via modified Lobene index scores 1-3.
* Medically free patients

Exclusion Criteria:

* Stains other than black.
* Patients on antibiotic treatment or any other medication for the last 2 weeks.
* Patients allergic to prophylaxis powder.
* Parents refusing to participate

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
chromogenic bacterial count before and after probiotic application | two weeks
  bacterial count

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry .Ain shams university, Cairo, Egypt